CLINICAL TRIAL: NCT04087876
Title: Expanded Access Use of Derazantinib for Patients With Locally Advanced, Inoperable or Metastatic iCCA Harbouring FGFR Genomic Alterations
Brief Title: Expanded Access Use of Derazantinib for Advanced Intrahepatic Cholangiocarcinoma (iCCA) With FGFR Genomic Alterations
Status: No longer available | Type: Expanded Access
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: DZB-iCCA-EA
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; iCCA; Metastatic cholangiocarcinoma; FGFR genomic alteration; biliary cancer; bile duct cancer; liver cancer
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms; Bile Duct Neoplasms; Liver Neoplasms | interventions — derazantinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: derazantinib — derazantinib will be administered orally

SUMMARY:
Basilea provided expanded access to derazantinib for patients with locally advanced, inoperable or metastatic intrahepatic cholangiocarcinoma (iCCA) with FGFR genomic alterations on a patient by patient basis while clinical development of derazantinib was ongoing.

ELIGIBILITY:
The following inclusion criteria were applied:

* all other treatment options had been exhausted
* patient was ineligible for any ongoing trials or was geographically inaccessible to trials including a trial with derazantinib
* there was a reason to believe that the potential benefit of receiving derazantinib outweighs the risk of treatment with an investigational drug product
* patient was willing and able to provide written informed consent
* if applicable, regulatory approval by the appropriate jurisdiction was obtained

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Häckl, MD, Study Director — Basilea Pharmaceutica International Ltd

REFERENCES:
- See also: Basilea Website — https://www.basilea.com/